CLINICAL TRIAL: NCT03869892
Title: An Open-label, Randomised, Phase III Study cOmparing trifLuridine/Tipiracil (S 95005) in Combination With Bevacizumab to Capecitabine in Combination With Bevacizumab in firST-line Treatment of Patients With metastatIC Colorectal Cancer Who Are Not candidatE for Intensive Therapy (SOLSTICE Study)
Brief Title: Phase III Study in First-line Treatment of Patients With Metastatic Colorectal Cancer Who Are Not Candidate for Intensive Therapy.
Acronym: SOLSTICE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL3-95005-006; 2017-004059-22 (EudraCT Number); U1111-1206-3198 (Other: UTN)
Record Dates: First submitted 2018-02-23; First posted 2019-03-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic; Cancer; Colorectal; Colorectal Cancer; Colon; Rectum; Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Neoplasms | interventions — Trifluridine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- S95005 + Bevacizumab (Experimental)
  Interventions: Drug: Trifluridine/tipiracil hydrochloride (S95005); Biological: Bevacizumab experimental
- Capecitabine + Bevacizumab (Active Comparator)
  Interventions: Drug: Capecitabine; Biological: Bevacizumab control

INTERVENTIONS:
Drug: Trifluridine/tipiracil hydrochloride (S95005) — Film-coated tablets of S 95005 (35 mg/m²/dose) will be administered orally twice a day (BID), within 1 hour after completion of morning and evening meals, 5 days on/2 days off, over 2 weeks, followed by a 14-day rest; This treatment cycle will be repeated every 4 weeks.
  Arms: S95005 + Bevacizumab
Drug: Capecitabine — Film-coated tablets, Capecitabine (1250 mg/m²/dose) will be administered orally BID on Days 1-14 of each cycle. This treatment cycle will be repeated every 3 weeks.
  Arms: Capecitabine + Bevacizumab
Biological: Bevacizumab experimental — Concentrate for solution for infusion, Bevacizumab (5 mg/kg, IV) administered every 2 weeks (Day 1 and Day 15). This treatment cycle will be repeated every 4 weeks.
  Arms: S95005 + Bevacizumab
Biological: Bevacizumab control — Concentrate for solution for infusion, Bevacizumab (7.5 mg/kg, IV) will be administered on Day 1 of each cycle.This treatment cycle will be repeated every 3 weeks.
  Arms: Capecitabine + Bevacizumab

SUMMARY:
The main purpose of this study is to demonstrate the superiority of S 95005 in combination with bevacizumab over capecitabine in combination with bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Has definitive histologically confirmed adenocarcinoma of the colon or rectum (all other histological types are excluded). Primary tumour localisation must be known.
2. RAS status based on local biological assessment of tumour biopsy must be available. If RAS status is not available at the time of randomisation, tumour biopsy must be available for RAS status determination (based on local biological assessment).
3. Patient is not a candidate for standard full dose combination chemotherapy with irinotecan or oxaliplatin
4. Patient is not a candidate for curative resection of metastatic lesions.
5. No previous systemic anticancer therapy for unresectable metastatic colorectal cancer.
6. ECOG (Eastern Cooperative Oncology Group) performance status ≤2.
7. Adequate organ function (renal, haematological, hepatic, coagulation) as described in the study protocol'

   Exclusion Criteria:
8. Pregnancy, breastfeeding or possibility of becoming pregnant during the study.
9. Participation in another interventional study within 4 weeks prior to the randomisation .
10. Patients who have not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy prior to the randomisation.
11. Symptomatic central nervous system metastases.
12. Major surgery within 4 weeks prior to the randomisation.

    Exclusion criteria related to S 95005 administration:
13. History of allergic reactions attributed to compounds of similar composition to S 95005 or any of its excipients.
14. Any contraindication present in the SmPC of trifluridine/tipiracil

    Exclusion criteria related to bevacizumab administration:
15. Any contraindication present in the SmPC of bevacizumab

    Exclusion criteria related to capecitabine administration:
16. Any contraindication present in the SmPC of capecitabine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 24 months
  Time elapsed between the randomization and the date of radiological tumour progression (according to RECIST 1.1) or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 8 years
  Time elapsed between the date of randomization and the date of death due to any cause.
Overall response rate (ORR) | Up to 8 years
  The proportion of patients with objective evidence of complete response (CR) or partial response (PR) according to RECIST 1.1 criteria and using investigator's tumour assessment.
Disease control rate (DCR) | Up to 8 years
  The proportion of patients with objective evidence of CR or PR or stable disease (SD) according to RECIST 1.1 criteria and using investigator's tumour assessment.
Duration of response (DoR) | Up to 8 years
  The time from the first documentation of response (CR or PR) to the first documentation of objective tumour progression or death due to any cause, whichever occurs first.
Time to treatment failure (TTF) | Up to 8 years
  The time from randomization to treatment discontinuation for any reason, including disease progression, treatment toxicity, patient preference, or death.
Incidence of Adverse Events (AEs) | Up to 8 years
Number of clinically significant changes to hematology, biochemistry, coagulation and urinalysis tests | Up to 8 years
Changes in ECOG performance status | Up to 8 years
Number of clinically significant changes to blood pressure, heart rate, body temperature and body weight | Up to 8 years
Number of clinically significant changes to 12-leads ECG parameters | Up to 8 years
Quality of life as assessed by EORTC QLQ-C30 | Up to 8 years
  European organization for research and treatment of cancer (EORTC) Quality of Life Questionnaire - Core Questionnaire (QLQ-C30) scores range from 0-100 and assess functional and symptom scores. For functional scores, a higher score represents an increase in functioning. For symptom scores, a higher score represents an increase in symptoms.
Quality of life as assessed by EQ-5D-5L | Up to 8 years
  The 5-level EQ-5D version questionnaire scores range from 5 to 25 with a higher score representing a worse health status.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, PhD, Principal Investigator — Medical Oncology departement Saint-Antoine hospital (Paris France 75012)
Locations (190):
- Argentina (10):
  - Centro de Oncología e Investigación de Buenos Aires COIBA, Berazategui
  - Hospital de Gastroenterología Dr. Carlos Borino Udaondo Oncology Unit, Buenos Aires
  - Fundación Favaloro Oncology Unit, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - Hospital Universitario CEMIC Servicio de Oncología, Unidad de tumores gastrointestinales, Buenos Aires
  - Centro Oncológico Riojano Integral CORI Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - Fundación COIR Centro Oncológico de Interación Regional, Mendoza
  - Centro Médico San Roque, San Miguel de Tucumán
  - Instituto de Oncología de Rosario, Santa Fe
  - ISIS Centro especializado, Santa Fe
- Australia (6):
  - Blacktown Hospital Cancer and Haematology Centre, Blacktown
  - Frankston Private Peninsula and Southeast Oncology Group, Frankston
  - Lake Macquarie Private Hospital, Gateshead
  - St George Hospital St George Hospital Cancer Care Centre, Kogarah
  - Adventist HealthCare Integrated Cancer Centre, Wahroonga
  - Southern Medical Day Care Centre, Wollongong
- Austria (6):
  - Med. Universität Graz Klinische Abteilung für Onkologie, Graz
  - Medizinische Universität Innsbruck Univ.-Klinik für Innere Medizin V, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern Interne I, Linz
  - Landeskrankenhaus (SALK) Universitätsklinik für Innere Medizin III (SALK), Salzburg
  - Universitätsklinikum St. Pölten Klinische Abteilung für Innere Medizin I, Sankt Pölten
  - Allgemeines Krankenhaus - Universitätskliniken Klinische Abteilung für Onkologie, Vienna
- Brazil (10):
  - Hospital do Câncer de Barretos - Fundação Pio XII Unidade de Pesquisa Clínica, Barretos
  - Cenantron - Clinica, Belo Horizonte
  - Sirio Libanes DF - Centro de Oncologia de Braslia do Sirio- Centro Intergrado de Pesquisa, Brasília
  - Centro de Pesquisa Hospital de Caridade de Ijuí Unidade de Pesquisa Clínica, Ijuí
  - Hospital Mae de Deus Oncologia, Porto Alegre
  - Hospital São Rafael Centro Intergrado de Pesquisa, Salvador
  - CEPHO - Centro de Estudos e Pesquisas em Hematologia e Oncol Centro Intergrado de Pesquisa, Santo André
  - Hospital de Base Centro Integrado de Pesquisa, São José do Rio Preto
  - ICESP - Instituto do Câncer do Estado de São Paulo Centro Integrado de Pesquisa, São Paulo
  - Hospital A C Camargo Unidade de Pesquisa Clinica, São Paulo
- Bulgaria (9):
  - "Complex oncology center - Burgas" EOOD Department of medical oncology, Burgas
  - "Multiprofile hosp. for active treatmen Dr. Tota Venkova" AD Department of medical oncology, Gabrovo
  - "Complex oncology center - Plovdiv" EOOD, IInd base Dpt. of Med. oncology and onc. diseases in gastroenterology, Plovdiv
  - "Medical Center Nadezhda Clinical" EOOD Medical Oncology Department, Sofia
  - "UMHAT Sv. Ivan Rilski" EAD Clinic of clinical hematology, Dpt. of medical oncology, Sofia
  - MHAT Serdika EOOD Department of Medical Oncology, Sofia
  - Spec. hospital for active treatment of oncology dis. EOOD Department of medical oncology and palliative care, Sofia
  - SHAT of oncology diseases Dr. Marko Antonov Markov" EOOD Department of medical oncology and palliative therapy, Varna
  - "Complex Ongology Center - Vratsa" EOOD Department of Medical oncology, Vratsa
- Czechia (5):
  - Masarykuv onkologicky ustav Klinika komplexni onkologicke pece, Brno
  - Fakultni nemocnice Ostrava Klinika onkologicka, Ostrava
  - Vseobecna fakultni nemocnice Onkologicka klinika VFN a 1. LF UK, Prague
  - Thomayerova nemocnice Onkologicka klinika 1. LF UK a TN, Prague
  - Fakultni nemocnice Olomouc Onkologicka klinika, Prague
- Denmark (4):
  - Aalborg Universitetshospital, Syd Onkologisk Afdelin, Aalborg
  - Rigshospitalet Onkologisk Klinik, Copenhagen
  - Regionshospitalet Herning, Hospitalsenheden Vest Onkologisk Afdeling, Herning
  - Odense Universitetshospital Onkologisk Afdeling R, Odense
- Estonia (3):
  - East Tallinn Central Hospital Center of Oncology, Tallinn
  - North Estonia Medical Centre Foundation Oncology and Haematology clinic, Tallinn
  - Tartu University Hospital, Hematology - Oncology clinic, Radiotherapy and oncological therapy, Tartu
- France (10):
  - Institut Sainte Catherine, Avignon
  - CHU Jean Minjoz Service d'oncologie médicale, Besançon
  - CHU Morvan Institut de Cancérologie et d'Hématologie, Brest
  - Hopital Privé Jean Mermoz Service de Gastro entérologie et d'Oncologie médicale, Lyon
  - Hôpital Nord Franche-Comté - Site du Mittan Service d'oncologie médicale, Montbéliard
  - Centre Antoine Lacassagne Dpt d'Oncologie Médicale, Nice
  - Hôpital Saint-Antoine Service d'Oncologie Médicale, Paris
  - Hôpital Européen Georges Pompidou Oncologie Hépatogastroenterologie-oncologie digestive, Paris
  - Hopital Haut-Leveque Hepato-gastroenterologie et oncologie digestive, Pessac
  - CHU Toulouse Rangueil Oncologie médicale digestive, Toulouse
- Germany (3):
  - Onkologische Schwerpunktpraxis Kurfuerstendamm, Berlin
  - Lübecker Onkologische Schwerpunktpraxis im Hochschulstadttei, Lübeck
  - Klinikum der Universität München Campus Großhadern, Medizinische Klinik und Poliklinik III, München
- Hungary (16):
  - Magyar Honvedseg Egeszsegugyi Kozpont Onkologiai Osztaly, Budapest
  - Semmelweis University Radiology and Oncotherapy Clinic, Budapest
  - Del-Pesti Centrumkh-Orsz. Hematologiai es Infektologiai Int. Szent Laszlo Telephely, Budapest
  - Szent Imre Egyetem Oktatokorhaz Klinikai Onkologia, Budapest
  - Orszagos Onkologiai Intezet "B" Belgyogyaszati-Onkologiai O. Es Klin. Farmakologiai O., Budapest
  - Uzsoki Utcai Korhaz Onkoradiologiai Osztaly, Budapest
  - Debreceni Egyetem Orvos es Egeszsegtudomanyi Centrum Onkologiai Intezet, Debrecen
  - Petz Aladar Megyei Oktato Korhaz Onkoradiologiai Osztaly, Győr
  - Bekes Megyei Kozponti Korhaz, Gyula
  - Bacs-Kiskun Megyei Korhaz Onkoradiologiai Kozpont, Kecskemét
  - Szabolcs-Szatmar-Bereg Megyei Korhazak Onkoradiologiai Osztaly, Nyíregyháza
  - Pecsi Tudomanyegyetem, Klinikai Kozpont Onkoterapias Intezet, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kp. Onkoterápiás Klinika, Szeged
  - JNSZ Megyei Hetenyi Geza Korhaz es Rendelointezet Megyei Onkologiai Centrum, Szolnok
  - Markusovsky Egyetemi Oktatokorhaz Onkoradiologiai Osztaly, Szombathely
  - Zala Megyei Korhaz Onkologiai osztaly, Zalaegerszeg
- Ireland (3):
  - Bon Secours Hospital, Cork
  - Cork University Hospital Department of Medical Oncology, Cork
  - The Adelaide and Meath Hospital, Dublin
- Italy (11):
  - Azienda Policlinico Universitaria - Presidio Monserrato Oncologia Medica, Cagliari
  - Azienda Socio Sanitaria Territoriale di Cremona ONCOLOGIA, Cremona
  - Istituto Nazionale Tumori I.R.C.C.S "Fondazione G. Pascale" Struttura Complessa di Oncologia Medica Addominale, Napoli
  - Istituto Oncologico Veneto IOV - IRCCS Unità Operativa Complessa Oncologia Medica 1, Padua
  - A.O.U. Pisana-Ospedale Santa Chiara U.O. di Oncologia Medica 2, Pisa
  - Ospedale San Carlo U.O. Oncologia Medica, Potenza
  - Arcispedale Santa Maria Nuova Unità di Oncologia, Reggio Emilia
  - Policlinico Universitario Campus Biomedico UOC di Oncologia Medica, Roma
  - Istituto Clinico Humanitas I.R.C.C.S Dipartimento di Oncologia Medica ed Ematologia, Rozzano (MI)
  - IRCSS Casa Sollievo della Sofferenza Dipartimento Onco-Ematologia, San Giovanni Rotondo
  - Ospedale S. Bortolo -ULSS8 Berica Distretto Est U.O. ONCOLOGIA, Vicenza
- Latvia (2):
  - P. Stradins Clinical University Hospital, Riga
  - Riga East Univerity Hospital Oncology Centre of Latvia, Riga
- Lithuania (4):
  - Oncology Hospital, Branch of Hospital of Lithuanian Uni. of Health Sciences Kauno klinikos, Kaunas
  - Hospital of Lithuania Univ of Health Sciences Kauno klinikos Oncology Institute, Kaunas
  - Klaipeda University hospital, Klaipėda
  - National Cancer Institute, Vilnius
- Netherlands (6):
  - Rijnstate Oncologie, Arnhem
  - Albert Schweitzer Ziekenhuis Interne Geneeskunde, Dordrecht
  - Catharina Ziekenhuis Interne Gesneeskunde/Oncologie, Eindhoven
  - Ikazia Ziekenhuis Oncologie, Rotterdam
  - ETZ Elisabeth Interne Geneeskunde, Tilburg
  - Bernhoven Interne Geneeskunde, Uden
- Poland (8):
  - Bialostockie Centrum Onkologii im Marii Curie-Sklodowskiej Oddzial Onkologii Klinicznej im Dr Ewy Pileckiej z pododdzialem Chemioterapii Dziennej, Bialystok
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii i Radioterapii, Gdansk
  - Przychodnia Lekarska "KOMED", Konin
  - M. Kopernika Provincial Hospital Oddzial Chemioterapii Nowotworow, Lodz
  - SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii Oddzial Kliniczny Onkologii i Immunoonkologii, Olsztyn
  - Opolskie Centrum Onkologii im. Tadeusza Koszarowskiego Oddzial Onkologii Klinicznej, Opole
  - Wielkopolskie Centrum Onkologii im Marii Sklodowskiej-Curie Oddzial Chemioterapii, Poznan
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej Tomaszów Mazowiecki II Sp. z o.o., Pododdzial Chemioterapi, Tomaszów Mazowiecki
- Portugal (5):
  - Hospital Garcia de Orta Serviço de Oncologia Médica, Almada
  - Centro Hospitalar e Universitário de Coimbra - CHUC Unidade de Inovação e Desenvolvimento (UID), Coimbra
  - Centro Hospitalar Lisboa Norte, Hospital de Santa Maria Serviço de Oncologia Médica, Lisbon
  - Hospital Beatriz Ângelo Serviço de oncologia medic, Loures
  - Instituto Português de Oncologia do Porto FG, EPE -IPO Porto Medical Oncology Dept., Porto
- Romania (8):
  - Institutul Oncologic "Prof Alexandru Trestioreanu" Busuresti Sectia Oncologie Medicala I, Bucharest
  - Spitalul Clinic "Coltea" Sectia Oncologie Medicala, Bucharest
  - Institutul Oncologic "Prof. Dr. I. Chiricuta" Cluj Napoca Oncologie Medicala, Cluj-Napoca
  - Centrul de Oncologie Sf Nectarie Oncology Department, Craiova
  - S.C Oncolab S.R.L Sectia Oncologie Medicala, Craiova
  - Institutul Regional de Oncologie Iasi Clinica de Oncologie Medicala, Iași
  - Spitalul Clinic Judetean de Urgenta Sibiu Sectia Oncologie Medicala, Sibiu
  - S.C ONCOMED S.R.L Departament Oncologie Medicala, Timișoara
- Russia (17):
  - Arkhangelsk Clinical Oncology Dispensary chemotherapy department, Arkhangelsk
  - Clinical Oncology Dispensary No.1 Chemotherapy Department, Krasnodar
  - Kursk Regional Clinical Oncology Dispensary Oncology Department, Kursk
  - Russian Cancer Research Center n.a. NN Blokhin Clinical Pharmacology and Chemotherapy, Moscow
  - University Headache Clinic Outpatient oncology clinic, Moscow
  - Moscow City Oncology Hospital # 62 chemotherapy department, Moscow
  - Omsk Clinical Oncologic Dispensary Chemotherapy, Omsk
  - Pyatigorsk Interdistrict Oncology Dispensary Chemotherapy department, Pyatigorsk
  - Rostov Research Institute of Oncology Chemotherapy department, Rostov-on-Don
  - Regional Clinical Oncology Dispensary, Ryazan
  - Scientific Centre for Specialized Medical Care (oncological) Chemotherapy, Saint Petersburg
  - National Medical Research Center of Oncology N.N. Petrova, Saint Petersburg
  - Saint Petersburg City Oncology Clilnic, Saint Petersburg
  - Multidisciplinary clinic "Reaviz", Samara
  - Oncology Dispensary No.2, Sochi
  - State Research Institution of Oncology of Tomsk Chemotherapy, Tomsk
  - SBIH of YR "Clinical oncology hospital" chemotherapy department, Yaroslavl
- Slovakia (2):
  - Narodny onkologicky ustav Oddelenie klinickej onkologie, Bratislava
  - Vychodoslovensky onkologicky ustav Oddelenie klinickej onkologie, Košice
- Spain (15):
  - Hospital General Universitario Alicante Servicio de Oncología, Alicante
  - Hospital Germans Trias i Pujol Unidad de Investigación clínica (UIC) ICO-Oncología medica, Badalona
  - H. Valle de Hebrón Servicio de Oncología - (VHIR), Barcelona
  - Hospital de la Santa Creu I Sant Pau Oncología Medica, Barcelona
  - Hospital Uni. Reina Sofía - Hospital Provincial Departamento de Oncología Médica, Córdoba
  - INSTITUTO CATALAN DE ONCOLOGÍA - ICO Oncología Médica, L'Hospitalet de Llobregat
  - Hospital Unviersitario Gregorio Marañon Servicio de Oncología Médica, Madrid
  - Hospital Universitario Ramón y Cajal, Servicio de Oncologia Médica, Madrid
  - H. Clínico San Carlos Servicio de Oncología Médica, Madrid
  - HOSPITAL 12 DE OCTUBRE Servicio Oncología Médica, Madrid
  - H. Universitario La Paz Oncología Médica, Madrid
  - Hospital Universitario Marqués de Valdecilla Oncología médica, Santander
  - H.Virgen Del Rocio, Seville
  - Hospital Quirónsalud Valencia Servicio de Oncología Médica, Valencia
  - Hospital Universitario Miguel Servet Servicio de Oncología, Zaragoza
- Sweden (5):
  - Falu Lasarett Onkologmottagningen, Falun
  - Lanssjukhuset Ryhov Onkologiska kliniken, Jönköping
  - Universitetssjukhuset Orebro, Örebro
  - Karolinska University Hospital, Solna Studiebehandlingsenheten, B8:09, Solna
  - Norrlands Universitetssjukhus Cancercentrum Umea, Umeå
- Ukraine (11):
  - Cherkasy Regional Oncological Dispensary Regional Clinical Oncological Centre, Cherkasy
  - Dnipro Regional Oncology Dispensary, Dnipro
  - MI "Dnipropetrovsk City Multi-field Clinical Hospital #4" Department of Oncology, Dnipro
  - Institute of Medical Radiology of S.P. Grygoryev of AMS UKR, Kharkiv
  - National Institute of Cancer Abdominal Oncology Department, Kyiv
  - Kyiv City Clinical Oncology Centre Chemotherapy Department #2, Kyiv
  - Municipal Institution of Kyiv Regional Council "Kyiv Regional Clinical Hospital", proctology department, Kyiv
  - Lviv Regional Oncology Center Chemotherapy department, Lviv
  - Odesa Regional Oncology Dispensary Day patient Department, Odesa
  - Podillia Regional Oncology Centre Chemotherapy Department, Vinnytsia
  - Regional Clinical Oncological Dispensary Department of Oncology, Zaporizhzhya
- United Kingdom (11):
  - Aberdeen Royal Infirmary Oncology Department, Aberdeen
  - University Hospitals Bristol Bristol Haematology & Oncology Centre, Bristol
  - St James's University Hospital, Leeds
  - Leicester Royal Infirmary The HOPE Clinical Trials Unit, Leicester
  - Royal Marsden Hospital Department of Medicine, London
  - Hammersmith Hospital Gary Weston Centre, London
  - Sarah Cannon Research Institute UK Clinical Trials, London
  - Imperial Healthcare NHS Trust Charing Cross Hospital, London
  - Christie Hospital NHS Foundation Trust GI & Endocrine, Manchester
  - Glan Clwyd Hospital North Wales Cancer Treatment Centre, Rhyl
  - Royal Marsden Hospital Department of Medicine, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Andre T, Falcone A, Shparyk Y, Moiseenko F, Polo-Marques E, Csoszi T, Campos-Bragagnoli A, Liposits G, Chmielowska E, Aubel P, Martin L, Fougeray R, Amellal N, Saunders MP. Trifluridine-tipiracil plus bevacizumab versus capecitabine plus bevacizumab as first-line treatment for patients with metastatic colorectal cancer ineligible for intensive therapy (SOLSTICE): a randomised, open-label phase 3 study. Lancet Gastroenterol Hepatol. 2023 Feb;8(2):133-144. doi: 10.1016/S2468-1253(22)00334-X. Epub 2022 Dec 2. PMID 36470291
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: study-level clinical trial data — https://clinicaltrials.servier.com/